CLINICAL TRIAL: NCT04897256
Title: Mobility in Daily Life and Falls in Parkinson's Disease: Potential for Rehabilitation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Martina Mancini, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01HD100383 (NIH); R01HD100383 (NIH)
Record Dates: First submitted 2021-05-18; First posted 2021-05-21 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Investigators involved in measuring outcomes and analyzing the data, will remain blinded to the group that participants are assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TURN-IT group (Experimental): Participants in the treatment group will attend supervised, 1-hour classes, 3 times per week for 6 weeks, one-on-one with the same exercise trainer, overseen by a physical therapist investigator.
  Interventions: Behavioral: TURN-IT exercise program
- No Intervention Control Group (No Intervention): Participants in this group will be tested at baseline and 6 weeks later. They will go about their normal daily life during the 6 week period.

INTERVENTIONS:
Behavioral: TURN-IT exercise program — Based on the exercise motor learning principles, participants spend 10-15 minutes at each Exercise Station that focuses on particular constraints of turning ability. The stations will focus on important underlying aspects of turning, such as weight-shifting and increasing axial rotation during functional turning tasks. Each station will be progressed across levels to make more challenging (such as adding a dual task). Initially participants will be supported in an overhead body-weight support system (ZeroG) to allow them to practice challenging exercises without the risk of falling.
  Arms: TURN-IT group

SUMMARY:
The goal of this intervention is to explore the effectiveness of a Turning Intervention (TURN-IT) to improve quality of turning in participants with Parkinson's Disease (PD). An unique exercise program has been developed - TURN-IT - in which participants practice exercises that focus on physiological constraints that impair turning ability, such as axial rigidity, narrow base of support, bradykinesia, and inflexible set-shifting. The 60 participants with PD and a history of falls in the previous 12 months, will be randomized into a 6-week, 3x/week, one-on-one TURN-IT group or No-Intervention Control group. This pilot intervention study will determine the number of subjects needed for a future clinical trial and will determine the sensitivity to change with rehabilitation our daily-life turning quality measures (such as, mean and variability of number of steps to turn, turn amplitude, turn velocity). The investigators predict that the TURN-IT program will improve turning in daily life enough to justify a larger clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of idiopathic PD from movement disorders neurologist with the United Kingdom Brain Bank criteria of bradykinesia with 1 or more of the following - rest tremor, rigidity, and balance problems not from visual, vestibular, cerebellar or proprioceptive conditions
2. Responsive to levodopa
3. Hoehn & Yahr stages II-IV
4. Age range 55-85 years old
5. self-report of one or more falls in past 12 months
6. willing and able to attend exercise intervention sessions at OHSU campus, and also refrain from changes in anti-parkinson medications and exercise levels.

Exclusion Criteria:

1. Major musculoskeletal or neurological disorders, structural brain disease, epilepsy, acute illness or health history, other than PD
2. no medical condition that precludes exercise
3. MoCA ≤ 21 or inability to follow directions
4. excessive use of alcohol or recreational drugs
5. recent change in medication
6. inability to stand and walk for 2 minutes without an assistive device

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2021-09-13 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in variability in number of steps to complete a turn | 6 weeks
  Coefficient of variation in the number of steps in a turn, averaged from daily monitoring

SECONDARY OUTCOMES:
Change in Falls Efficacy Scale International | 6 weeks
  A 16 item self-administered questionnaire to assess fear of falling. Score range 16-64 with higher score indicating more fear of falling
Change in prospective fall rate | 52 weeks
  Number of prospective falls recorded for 12 months starting from the end of intervention
Change in patient global impression of change | 6 weeks
  Question of participant's rating of mobility. Score range from 1-7 with 1-3 indicating improvement, 4 no change, and 5-7 worsening of mobility
Change in number of steps to complete a turn | 6 weeks
  Number of steps in a turning averaged from daily monitoring
Change in turn peak velocity | 6 weeks
  Peak velocity of turns averaged from daily monitoring
Change in turn angle amplitude | 6 weeks
  Peak size of turn angles averaged from daily monitoring
Change in turn duration | 6 weeks
  Time to complete turns averaged from daily monitoring
Change in turn trunk jerk | 6 weeks
  A measure of smoothness of turning; the rate of change of acceleration during a turn averaged from daily monitoring
Change in variability of double-support time | 6 weeks
  Coefficient of variation in time of double-support phase
Change in lateral trunk range | 6 weeks
  range of motion in the trunk during walking, in the lateral direction

OTHER OUTCOMES:
Change in mini-Balance Evaluation Systems Test | 6 weeks
  Clinical measure of four balance domains-anticipatory, reactive, sensory, and dynamic gait. Scores range from 0-28 with higher scores indicating worse balance
Change in clinical global impression of change | 6 weeks
  Question of clinician's rating of participant mobility. Score range from 1-7 with 1-3 indicating improvement, 4 no change, and 5-7 worsening of mobility.
Change in Parkinson's Disease Questionnaire-39 | 6 weeks
  A 39 item self-report questionnaire to assess Parkinson's disease specific health related quality in eight domains of quality of life. Each item scores from 0 (never) to 4 (always). Sub-scale scores and a Parkinson's Disease summary index (PDSI; sum of eight subsections/8) representing the global health-related quality of life will be calculated, with higher scores representing worse quality of life
Change in Unified Parkinson's Disease Rating Scale, Part III | 6 weeks
  A clinical scale to assess severity of motor symptoms in Parkinson's disease. Each item is scored 0 (normal) to 4 (severe) with a score range from 0-132
Change in Activities-Specific Balance Confidence Scale | 6 weeks
  A 16-item self-report scale that participants rate their confidence in performing daily activities. Score range from 0-100% with 0% meaning no confidence and 100% completely confident
Change in stride velocity | 6 weeks
  Stride velocity during straight walking averaged from daily monitoring
Change in stride length | 6 weeks
  Stride length during straight walking averaged from daily monitoring
Change in cadence | 6 weeks
  The number of straight walking steps taken per minute averaged from daily monitoring
Change in double support time | 6 weeks
  The amount of time both feet were on the ground together during straight walking averaged from daily monitoring
Change in angle of foot at heel strike | 6 weeks
  The angle between the foot and the ground at heel strike during straight walking averaged from daily monitoring
Change in variability of angle of foot at heel strike | 6 weeks
  Coefficient of variation of the angle between the foot and the ground at heel strike during straight walking averaged from daily monitoring
Change in number of turns per hour | 6 weeks
  The average number of turns per hour measured during daily monitoring
Change in number of bouts of walking and steps per day | 6 weeks
  The average number of walking bouts and number of steps per day, measured during daily monitoring
Change in duration of longest walking bout per day | 6 weeks
  The longest bout of straight walking per day averaged from daily monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Fay Horak, PhD, PT, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request, we can share de-identified data related to study outcomes measures.
Supporting Information: Study Protocol, SAP
Time Frame: Data would be available 6 months after the end of data collection. Data will be stored in our laboratory data repository and so will be available indefinitely.
Access Criteria: Data will not be stored on a public website, however researchers may contact us for access to the data. We will send data electronically via a secure server.

REFERENCES:
- [Derived] King LA, Carlson-Kuhta P, Wilhelm JL, Lapidus JA, Dale ML, Talman LS, Barlow N, Mancini M, Horak FB. TURN-IT: a novel turning intervention program to improve quality of turning in daily life in people with Parkinson's disease. BMC Neurol. 2022 Nov 28;22(1):442. doi: 10.1186/s12883-022-02934-5. PMID 36443737